CLINICAL TRIAL: NCT05765578
Title: DisCOVEries 2 - An Observational Study to Evaluate the Immunogenicity of mRNA COVID-19 Bivalent Vaccines (Original and Omicron BA.4/BA.5) and 2023 Updated mRNA COVID-19 Vaccines (XBB.1.5)
Brief Title: An Observational Study of Moderna COVID-19 Bivalent Vaccines (Original and Omicron BA.4/BA.5) and 2023 Updated mRNA COVID-19 Vaccines (XBB.1.5)
Status: Completed | Type: Observational
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: mRNA-1273-P922
Record Dates: First submitted 2023-03-09; First posted 2023-03-13 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: COVID-19
Keywords: Immunogenicity; Moderna; mRNA-1273; Omicron; Vaccines
MeSH Terms: conditions — COVID-19 | interventions — 2019-nCoV Vaccine mRNA-1273; BNT162 Vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Serum from blood samples will be used for binding antibody testing.

GROUPS / COHORTS (4):
- Moderna-Only Vaccine/Booster Series (MMMM Group): Individuals who previously received Moderna COVID-19 vaccines in both primary series and first booster and a bivalent booster against Omicron BA.4/5 as the second booster dose (Moderna mRNA1273.222).
  Interventions: Biological: Moderna COVID-19 Vaccine; Biological: Moderna mRNA1273.222 Booster
- Pfizer-Only Vaccine/Booster Series (PPPP Group): Individuals who previously received Pfizer COVID-19 vaccines in both primary series and first booster and a bivalent booster against Omicron BA.4/5 as the second booster dose (Pfizer-BNT 162b2 bivalent booster).
  Interventions: Biological: Pfizer COVID-19 Vaccine
- Moderna mRNA COVID-19 updated vaccine (XBB.1.5): Comparison Group: Individuals who received Moderna 2023 updated COVID-19 vaccine (XBB.1.5).
  Interventions: Biological: Moderna 2023 Updated COVID-19 vaccine (XBB.1.5)
- Pfizer-BioNTech COVID-19 updated vaccine (XBB.1.5): Reference Group: Individuals who received Pfizer 2023 updated COVID-19 vaccine (XBB.1.5).
  Interventions: Biological: Pfizer 2023 Updated COVID-19 vaccine (XBB.1.5)

INTERVENTIONS:
Biological: Moderna COVID-19 Vaccine — Sterile liquid for injection. Intervention not administered through this study.
  Groups: Moderna-Only Vaccine/Booster Series (MMMM Group)
Biological: Moderna mRNA1273.222 Booster — Sterile liquid for injection. Intervention not administered through this study.
  Groups: Moderna-Only Vaccine/Booster Series (MMMM Group)
Biological: Pfizer COVID-19 Vaccine — Sterile liquid for injection. Intervention not administered through this study.
  Groups: Pfizer-Only Vaccine/Booster Series (PPPP Group)
Biological: Moderna 2023 Updated COVID-19 vaccine (XBB.1.5) — Sterile liquid for injection. Intervention not administered through this study.
  Groups: Moderna mRNA COVID-19 updated vaccine (XBB.1.5): Comparison Group
Biological: Pfizer 2023 Updated COVID-19 vaccine (XBB.1.5) — Sterile liquid for injection. Intervention not administered through this study.
  Groups: Pfizer-BioNTech COVID-19 updated vaccine (XBB.1.5): Reference Group

SUMMARY:
The goal of this observational study is to analyze binding antibody levels in adults in the United States (US) after receiving coronavirus disease 2019 (COVID-19) bivalent boosters (original and omicron BA.4/5) and updated COVID-19 vaccines (XBB.1.5).

ELIGIBILITY:
Inclusion Criteria:

* Lives in the continental United States (US).
* Speaks, reads, and understands English.
* Is willing and able to submit vaccination card photo(s) or vaccination records.
* Is willing and able to self-collect capillary blood during the study period via an at-home whole-blood collection device.
* Is fully vaccinated against COVID-19 per protocol specified criteria.

Exclusion Criteria:

* Has been diagnosed with significant cognitive impairment or dementia.
* Is pregnant or planning to become pregnant during the study period.
* Primary mailing address is a Post Office box, Army Post Office, Fleet Post Office, or Diplomatic Post Office address.
* Currently lives in a US military base located overseas, or US territories (Puerto Rico, US Virgin Islands, Guam, Northern Mariana Island, or American Samoa).
* Is currently participating in a COVID-19 vaccine clinical trial.
* Is currently receiving chemotherapy or has received chemotherapy in the past 6 months.
* Is currently taking steroids, such as prednisone, for any condition.
* Has been diagnosed with and taking immunosuppressants for rheumatoid arthritis, lupus or multiple sclerosis.
* Has received an organ transplant.
* Is currently undergoing dialysis of any kind (for example, hemodialysis or chronic ambulatory dialysis) for kidney disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants who have received the COVID-19 vaccine(s) and booster.
Sampling Method: Non-Probability Sample
Enrollment: 1713 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
Geometric Mean Titer (GMT) of Serum Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Binding Antibody Titers Against Omicron BA.4/5 at Day 29 Between MMMM Group and PPPP Group | Day 29
GMT of SARS-CoV-2 Binding Antibody Titers Against Omicron BA.4/5 at Day 91 Between MMMM Group and PPPP Group | Day 91
GMT of SARS-CoV-2 Binding Antibody Titers Against Omicron BA.4/5 at Day 181 Between MMMM Group and PPPP Group | Day 181
Geometric Mean Ratio (GMR) of GMT of Serum SARS-CoV-2 Binding Antibody Concentrations Against Omicron XBB.1 at Day 29 Between Moderna 2023 Updated COVID-19 vaccine (XBB.1.5) and Pfizer 2023 Updated COVID-19 vaccine (XBB.1.5) | Day 29
GMR of GMT of Serum SARS-CoV-2 Binding Antibody Concentrations Against Omicron XBB.1 at Day 91 Between Moderna 2023 Updated COVID-19 vaccine (XBB.1.5) and Pfizer 2023 Updated COVID-19 vaccine (XBB.1.5) | Day 91
GMR of GMT of Serum SARS-CoV-2 Binding Antibody Concentrations Against Omicron XBB.1 at Day 181 Between Moderna 2023 Updated COVID-19 vaccine (XBB.1.5) and Pfizer 2023 Updated COVID-19 vaccine (XBB.1.5) | Day 181

SECONDARY OUTCOMES:
GMT Against All Other Omicron Variants and Subvariants Between MMMM Group and PPPP Group | Day 29, Day 91, and Day 181
GMR of GMT Against All Other Omicron Variants and Subvariants Between Moderna 2023 Updated COVID-19 vaccine (XBB.1.5) and Pfizer 2023 Updated COVID-19 vaccine (XBB.1.5) | Day 29, Day 91, and Day 181

CONTACTS AND LOCATIONS:
Locations (1):
- Science37, Culver City, California, United States